CLINICAL TRIAL: NCT00527995
Title: Acute Effects of Sildenafil on Flow Mediated Dilatation and Cardiovascular Autonomic Nerve Function in Type 2 Diabetic Patients
Brief Title: Acute Effects of Sildenafil on Endothelial Function in People With Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Sildenafil_ED_2001
Record Dates: First submitted 2007-09-10; First posted 2007-09-11 (Estimated); Last update posted 2007-09-11 (Estimated); Status verified 2007-09

CONDITIONS: Type 2 Diabetes Mellitus; Endothelial Dysfunction
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sildenafil — Orally administered, Sildenafil 100mg, unique administration
  Other Names: Viagra

SUMMARY:
This is a double-blind, placebo-controlled, cross-over trial using a single dose of 100 mg sildenafil or placebo in 40 subjects with T2DM without known cardiovascular disease. Effects on haemodynamic parameters, flow mediated dilatation (FMD) in brachial artery, cardiovascular autonomic function tests, and spontaneous baroreflex sensitivity (BRS) were investigated.

ELIGIBILITY:
Inclusion Criteria:

* age 35-70
* type 2 diabetes mellitus
* impotence
* with and without hypertension, hypercholesteremia

Exclusion Criteria:

* patients with history of cardiovascular and malignant disease,
* advanced nephropathy (creatinine≥2.2mg/dl)
* hepatopathy (liver enzymes higher than the double of normal values)
* patients taking nitrates
* CHF: NYHA > II
* Stable angina: CCS > II

Ages: 35 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2001-08; Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Improvement of flow mediated dilatation of the brachial artery following a single dose of 100mg Sildenafil. | 60 minutes

SECONDARY OUTCOMES:
Change in hemodynamics and cardiovascular parasympathetic and sympathetic nerve function using time domain and frequency domain indexes of heart rate variability (HRV) and baroreflex sensitivity (BRS) following a single dose of 100mg Sildenafil. | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Alin Stirban, MD, Principal Investigator — Heart and Diabetes Center NRW; Dan Ziegler, MD, Study Director — German Diabetes Center Duesseldorf
Locations (1):
- German Diabetes Center, Düsseldorf, North Rhine-Westphalia, Germany